CLINICAL TRIAL: NCT03634670
Title: The Influence of Interdisciplinary Multimodal Pain Therapy on Cerebral Connectivity in Chronic Pain Patients
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: German Research Foundation (Other); Technical University of Munich, Center for Interdisciplinary Pain Medicine, Klinikum rechts der Isar (Unknown)
Responsible Party: Sponsor
Other Study IDs: 01/2018
Record Dates: First submitted 2018-05-14; First posted 2018-08-16 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Chronic Pain, Interdisciplinary Multimodal Pain Therapy, Electroencephalography, Functional Connectivity
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interdisciplinary multimodal pain therapy (IMPT) — The IMPT-program is provided in a specialized day-clinic setting over a period of 20 treatment days. There are two different treatment programs with either 5 days per week over a period of 4 weeks or 3 days per week over a period of 7 weeks. IMPT comprises individual pharmacotherapy evaluated in regular consultations with a physician as well as a structured physiotherapy and psychotherapy programs on group level and individual level. Group physiotherapy comprises exercise therapy, movement experience and relaxation techniques. Additionally individual physiotherapy is provided in two extra sessions focusing on the individual needs and problems of the patient. Group psychotherapy comprises educational contents (e.g. pathophysiology and biopsychosocial aspects of pain) as well as cognitive-behavioral-interventions e.g. regarding stress-management. Additionally individual psychotherapy is provided in four extra sessions focusing on the individual needs and problems of the patient.

SUMMARY:
Due to its high prevalence and the substantial individual and socio-economic burden chronic pain is a huge challenge for patients, physicians and the society. Using neuroimaging structural and functional alterations have been described in the brain of patients suffering from chronic pain (Apkarian, Hashmi et al. 2011, Baliki and Apkarian 2015). However, reproducibility and functional significance of these changes are only incompletely understood. For example it remains unclear, if these changes covariate with clinical parameters and if they can be influenced or reversed by appropriate therapy. Some of the structural and functional brain changes in chronic pain patients have been shown to be reversible using magnetic resonance imaging after successful interventional pain treatment (Seminowicz, Wideman et al. 2011) or cognitive-behavioral therapy (Seminowicz, Shpaner et al. 2013, Shpaner, Kelly et al. 2014). Interdisciplinary multimodal pain therapy (IMPT) as a biopsychosocial treatment approach comprising physiotherapy and psychotherapy in structured programs has been shown to be effective in alleviating chronic pain of different entities including those where interventional therapy options are lacking or have been unsuccessful (Kaiser, Treede et al. 2017). The present study aims to investigate the influence of a structured IMPT approach provided in a day-clinic program of 20 treatment days on the functional brain network structure in chronic pain patients. To this end, a graph-theory based analysis (Bullmore and Sporns 2009) will be applied to electroencephalography (EEG) resting-state data from 30 chronic pain patients before and after IMPT and results will be correlated with behavioral and clinical data. In this observational study chronic pain patients that have been screened for participation in IMPT as part of routine medical care are invited to participate in a baseline visit prior to participation and a follow-up visit 6 months after completion of the program.

This will add to a better understanding of the complex functional brain alterations in chronic pain and might contribute to identify neuronal markers or even predictors for therapeutic responses in multimodal pain treatments. Moreover, the broad availability and easy applicability of EEG-measurements might enable a wide therapeutic application of potential findings in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain (duration >6 months, not primary headache disease)
* Willing and able to comply with physical (e.g. able to get up from the floor without help) and psychological (e.g. motivation for behavioural change) requirements of the IMPT-day-clinic setting as assessed by a physician, psychologist and physiotherapist on a screening visit as part of routine medical care prior to participation
* Willing and able to sign informed consent for study participation

Exclusion Criteria:

* Recent change in chronic pain condition (e.g. surgery or injury within the last 3 months)
* Concomitant neurological or psychiatric disease apart from Depression (especially severe mental disorder or psychopathology)
* Regular (daily) intake of benzodiazepines
* Addiction problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All chronic pain patients eligible according to the inclusion and exclusion criteria (see eligibility criteria) participating in the IMPT-day-clinic programme of the Center for Interdisciplinary Pain Medicine at the Klinikum rechts der Isar of the Technische Universität München in the year 2018 are invited to voluntarily participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline visual analogue scale (VAS) ratings of pain intensity at 6 months | Measured at baseline and at 6 months post treatment
  Pain rating for average Pain intensity within the last 4 weeks on the VAS ranging from 0=no pain to 10=worst imaginable pain

SECONDARY OUTCOMES:
Change from baseline Pain related disability / Quality of life / Depression / Pain characteristics at 6 months | Measured at baseline and at 6 months post treatment
  Metrics assessed using the German Pain Questionnaire (Nagel, Gerbershagen et al. 2002), short-form McGill Pain Questionnaire (Melzack 1987), Beck Depression Inventory II (Beck et al 1986), painDETECT Questionnaire (Freynhagen et al 2006)

OTHER OUTCOMES:
Change from baseline functional cerebral connectivity as assessed by resting-state Electroencephalography (EEG) at 6 months | Measured at baseline and 6 months post treatment
  64-Channel-EEG resting state measurements and Graph-theory based analysis of frequency bands (gamma, beta, alpha, theta, delta) on sensor and source level including degree centrality, clustering coefficient, global efficiency, small-worldness, modularity und global hub disruption index

CONTACTS AND LOCATIONS:
Overall Officials: Markus Ploner, Professor, MD, Principal Investigator — Department of Neurology, Klinikum rechts der Isar, TUM
Locations (1):
- Department of Neurology, Center for Interdisciplinary Pain Medicine, Klinikum rechts der Isar, TUM, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Apkarian VA, Hashmi JA, Baliki MN. Pain and the brain: specificity and plasticity of the brain in clinical chronic pain. Pain. 2011 Mar;152(3 Suppl):S49-S64. doi: 10.1016/j.pain.2010.11.010. Epub 2010 Dec 13. PMID 21146929
- [Background] Baliki MN, Apkarian AV. Nociception, Pain, Negative Moods, and Behavior Selection. Neuron. 2015 Aug 5;87(3):474-91. doi: 10.1016/j.neuron.2015.06.005. PMID 26247858
- [Background] Bullmore E, Sporns O. Complex brain networks: graph theoretical analysis of structural and functional systems. Nat Rev Neurosci. 2009 Mar;10(3):186-98. doi: 10.1038/nrn2575. Epub 2009 Feb 4. PMID 19190637
- [Background] Kaiser U, Treede RD, Sabatowski R. Multimodal pain therapy in chronic noncancer pain-gold standard or need for further clarification? Pain. 2017 Oct;158(10):1853-1859. doi: 10.1097/j.pain.0000000000000902. No abstract available. PMID 28328572
- [Background] Nagel B, Gerbershagen HU, Lindena G, Pfingsten M. [Development and evaluation of the multidimensional German pain questionnaire]. Schmerz. 2002 Aug;16(4):263-70. doi: 10.1007/s00482-002-0162-1. German. PMID 12192435
- [Background] Seminowicz DA, Shpaner M, Keaser ML, Krauthamer GM, Mantegna J, Dumas JA, Newhouse PA, Filippi CG, Keefe FJ, Naylor MR. Cognitive-behavioral therapy increases prefrontal cortex gray matter in patients with chronic pain. J Pain. 2013 Dec;14(12):1573-84. doi: 10.1016/j.jpain.2013.07.020. Epub 2013 Oct 14. PMID 24135432
- [Background] Seminowicz DA, Wideman TH, Naso L, Hatami-Khoroushahi Z, Fallatah S, Ware MA, Jarzem P, Bushnell MC, Shir Y, Ouellet JA, Stone LS. Effective treatment of chronic low back pain in humans reverses abnormal brain anatomy and function. J Neurosci. 2011 May 18;31(20):7540-50. doi: 10.1523/JNEUROSCI.5280-10.2011. PMID 21593339
- [Background] Shpaner M, Kelly C, Lieberman G, Perelman H, Davis M, Keefe FJ, Naylor MR. Unlearning chronic pain: A randomized controlled trial to investigate changes in intrinsic brain connectivity following Cognitive Behavioral Therapy. Neuroimage Clin. 2014 Jul 23;5:365-76. doi: 10.1016/j.nicl.2014.07.008. eCollection 2014. PMID 26958466
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Beck, A.T., Steer, R.A., & Brown, G.K. (1996). Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation.
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Derived] Heitmann H, Gil Avila C, Nickel MM, Ta Dinh S, May ES, Tiemann L, Hohn VD, Tolle TR, Ploner M. Longitudinal resting-state electroencephalography in patients with chronic pain undergoing interdisciplinary multimodal pain therapy. Pain. 2022 Sep 1;163(9):e997-e1005. doi: 10.1097/j.pain.0000000000002565. Epub 2021 Dec 15. PMID 35050961